CLINICAL TRIAL: NCT01298050
Title: Refractory In and Out of Hospital Cardiac Arrest Treated With Extracorporeal Membrane Oxygenation. Observational, Single Centre, Prospective Study.
Brief Title: Refractory IHCA and OHCA Treated With ECMO
Acronym: SEAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milano Bicocca (Other)
Collaborators: Ospedale San Gerardo. S.S.U.E.M. 118 Brianza (Unknown); Ospedale San Gerardo. Terapia Intensiva Cardiochirurgica (Unknown)
Responsible Party: Roberto Fumagalli, University of Milano Bicocca
Other Study IDs: AOSG-TICCH-01-2011
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-07

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Extracorporeal Membrane Oxygenation: All patients have to start ECMO under CPR, by insertion of peripheral VA cannulas.
  Interventions: Procedure: ECMO

INTERVENTIONS:
Procedure: ECMO — Insertion of peripheral Veno-Arterious ECMO, subsequent therapeutic hypothermia

SUMMARY:
Extracorporeal membrane oxygenation (ECMO) support has been suggested to improve the survival rate in patients with refractory cardiac arrest (CA). Recent studies have also highlighted the potential early application of this method in improving the prognosis of prolonged cardiac arrest both for in hospital CA (INHCA) and out of hospital CA (OHCA). The rationale for use of ECMO in these patients is to optimize early perfusion of vital organs, curing the cause of CA and waiting for the recovery of the injured myocardium. The investigators have created a flow-chart to decide which patients are eligible. The aims of this study are to evaluate if, with this flow-chart, the investigators are able to detect which patients have more probability of survival.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-75 years old
* In and out of hospital Witnessed Cardiac Arrest
* No-flow time < 5 min. or VF,VT,TP as rhythm of presentation
* Low-flow time < 45 min.
* End Tidal CO2 > 10 after 20 min.of CPR

Exclusion Criteria:

* Comorbidities such:
* Terminal Malignancy
* Aortic Dissection
* Severe Cardiac Failure without transplant indication
* Severe Aortic Valve Failure
* Known Severe Peripheral arteriopathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults 18-75 years old, community sample
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
28 days survival | 28 days

SECONDARY OUTCOMES:
Neurologic recovery | 28 days
  Neurologic recovery defined as minimal neurologic impairment according to the Glasgow-Pittsburgh cerebral performance categories score ≤ 2.
Cardiac recovery | 28 days
  Measured by echocardiography
Six months survival with minimal neurologic impairment | 180 days
  survival with minimal neurologic impairment according to the Glasgow-Pittsburgh cerebral performance categories score ≤ 2.

CONTACTS AND LOCATIONS:
Overall Officials: Leonelllo Avalli, MD, Principal Investigator — Ospedale San Gerardo
Locations (1):
- San Gerardo Hospital, Monza, MB, Italy